CLINICAL TRIAL: NCT00245531
Title: Effects of Endocrine Health on the Cognitive Function of Men and Women Using Drugs: A Cross-sectional Investigation
Brief Title: Effects of Endocrine Health on Mental Performance of Men and Women Using Drugs
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Adrian S. Dobs, Professor of Medicine and Oncology, Johns Hopkins University
Other Study IDs: 05-01-12-04
Record Dates: First submitted 2005-10-25; First posted 2005-10-28 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Human Immunodeficiency Virus Positive or Negative
Keywords: endocrine abnormalities; cognitive performance
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- +IDU/+HIV or -HIV
- -IDU and -HIV (controls)

SUMMARY:
The purpose of this study is to understand the effects of decreased functioning of the testes or ovaries on mental performance in males and females using illicit drugs excluding marijuana.

DETAILED DESCRIPTION:
This research is being done to understand the effects of endocrine abnormalities, specifically hypogonadism (decreased functioning of the testes or ovaries) on cognitive (mental) performance in males and females using illicit drugs (excluding marijuana).

ELIGIBILITY:
Inclusion Criteria:

* Completed the 8th grade

Exclusion Criteria:

* Did not complete the 8th grade. Have a hormone problem for which you are taking medication e.g. testosterone or thyroid medicine, steroids, oral contraceptives, progesterone. Diagnosed with cancer. History of schizophrenia. Currently have or have been diagnosed in the past with meningitis or encephalitis.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: males and females 18-50 years old who have completed the 8th grade and are using drugs
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2004-08; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Cognitive function | 12 weeks
  Performance on visuospatial, fine motor and verbal tasks can be poor in hypogonadal populations of men and women. HIV+ and IDU+ populations often experience endocrine abnormalities such as hypogonadism. The goal of Study 1 is to determine if patterns of cognitive performance associated with hypogonadism generalize to IDU+, HIV+/HIV- populations. Furthermore, an attempt will be made to associate patterns of cognitive performance with specific endocrine measures, IDU status, HIV status and QOL measures. All published testing materials have been shown to provide good reliability.

SECONDARY OUTCOMES:
Gonadal hormones | 12 weeks
  Serum sex hormone measurements are reliable blood tests commonly used to evaluate gonadal function. Total testosterone, the most frequently used screening test for hypogonadism in men, is relatively inexpensive and reliable; free testosterone is loosely bound to albumin. Levels of LH and FSH will assist in discriminating between a central vs. primary hypogonadism. Estradiol is expected to correlate with testosterone levels in men, since testosterone is aromatized to estradiol in the adipocyte. Based on the literature, it is expected that men and women IDU+ will have centrally mediated (secondary hypogonadism) with decreases in serum FSH, LH, estradiol and androgens.

OTHER OUTCOMES:
Quality of life | 12 weeks
  We intend to examine associations between measures of QOL and the cognitive and endocrine measures described above.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian S Dobs, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, The Clinical Trials Unit, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Goldberg CS, Trachtenberg F, William Gaynor J, Mahle WT, Ravishankar C, Schwartz SM, Cnota JF, Ohye RG, Gongwer R, Taylor M, Paridon S, Frommelt PC, Afton K, Atz AM, Burns KM, Detterich JA, Hill KD, Cabrera AG, Lewis AB, Pizarro C, Shah A, Sharma B, Newburger JW; Pediatric Heart Network Investigators. Longitudinal Follow-Up of Children With HLHS and Association Between Norwood Shunt Type and Long-Term Outcomes: The SVR III Study. Circulation. 2023 Oct 24;148(17):1330-1339. doi: 10.1161/CIRCULATIONAHA.123.065192. Epub 2023 Oct 5. PMID 37795623
- [Derived] Zilbermint MF, Wisniewski AB, Xu X, Selnes OA, Dobs AS. Relationship between sex hormones and cognitive performance in men with substance use. Drug Alcohol Depend. 2013 Mar 1;128(3):250-4. doi: 10.1016/j.drugalcdep.2012.08.024. Epub 2012 Sep 26. PMID 23021515